CLINICAL TRIAL: NCT05949125
Title: Multicenter, Open-label, Phase 1 Study of Allo-RevCAR01-T-CD123 Consisting of Genetically Modified T Cells Carrying Reverse Chimeric Antigen Receptors (Allo RevCAR01 T) in Combination With CD123 Target Module (R-TM123) for the Treatment of Patients With Selected Hematologic Malignancies Positive for CD123
Brief Title: Phase 1 Study of Allo-RevCAR01-T-CD123 in Patients With Selected CD123 Positive Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AvenCell Europe GmbH (Industry)
Collaborators: Allucent (NL) BV (Unknown)
Responsible Party: Sponsor
Organization: AvenCell Therapeutics, Inc. (Industry)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVC-201-01; 2022-501797-19-00 (Other: EU CT Number)
Record Dates: First submitted 2023-06-23; First posted 2023-07-17 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia Refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: The initial dose escalation (Escalation 1) follows a BOIN comb design with 3 dose levels of Allo-RevCAR01-T and 3 dose levels of R-TM123 resulting in a maximum of 9 dose levels. Given 1 participant dose level cohorts, there will be an inherent stagger between each participant equivalent to the DLT window of 28 days. Dose escalation 1 is followed by a second escalation phase (Escalation 2), including three more R-TM123 dose levels, in combination with the maximum cell dose obtained during the escalation 1. The three additional dose levels will be investigated via a classical 3+3 design (three patients will be treated per dose cohort). If a DLT is observed, three more patients will be added to that dose level.
  After escalation, two randomized expansion cohorts (≥10 R/R AML patients each) will compare dose levels to define Phase 2 dosing. If one dose in escalation phase proves clearly superior, a non-randomized Phase 1b expansion with up to 20 patients at that dose may be initiated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allo-RevCAR01-T-CD123 treatment (Experimental): Following lymphodepleting therapy, R-TM123 will be administered as continuous infusion from Cycle 1 Day 1 and then will continue for 20 days. Allo-RevCAR01-T will be administered on Day 1.
  Participants who tolerate Cycle 1 of R-TM123 and Allo-RevCAR01-T without DLT and are not diagnosed with disease progression after Cycle 1, will be considered for consolidation cycles of 12 consecutive days each of continuous IV infusion of R-TM123 until relapse, unacceptable toxicity, potentially curative treatment option (alloHSCT), consent withdrawal, or maximum one year treatment time.
  Interventions: Other: Cyclophosphamide (Non-IMP, Lymphodepletion); Other: Fludarabine (Non-IMP, Lymphodepletion); Drug: R-TM123; Drug: Allo-RevCAR01-T

INTERVENTIONS:
Other: Cyclophosphamide (Non-IMP, Lymphodepletion) — Intravenous infusion over 3 days (d-5 to d-3)
Other: Fludarabine (Non-IMP, Lymphodepletion) — Intravenous infusion over 3 days (d-5 to d-3)
Drug: R-TM123 — Intravenous infusion over 20 days
  Other Names: R-TM123 is one component of the Allo-RevCAR01-T-CD123 treatment
Drug: Allo-RevCAR01-T — Allo-RevCAR01-T will be administered as IV infusion on Treatment day 1.
  Other Names: Allo-RevCAR01-T is one component of the Allo-RevCAR01-T-CD123 treatment

SUMMARY:
The Allo-RevCAR01-T-CD123 drug is a combination of a cellular component (Allo-RevCAR01-T) with a recombinant antibody derivative (R-TM123), which together form the active drug. The cellular component Allo-RevCAR01-T consists of an allogeneic human T-cell genetically multi-edited and expressing a reversed, universal chimeric antigen receptor (RevCAR) presenting an extracellular peptide epitope (RevCAR epitope). R-TM123 functions as a bridging module between Allo-RevCAR01-T and a CD123-expressing target cancer cell by selectively binding the RevCAR epitope and CD123.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants, age ≥18 years. 2. HLA type of participant must match at HLA B and C loci 3.

1. For Phase 1a escalation part of the trial Participants with CD123+ AML (defined as ≥20% of leukemic cells expressing CD123 at any point in the course of disease)

   (1) for whom all standard or life-extending therapies have failed and for whom no potentially curative therapies are available or who are intolerant to such therapies.
2. For Phase 1b expansion part of the trial (Phase 1b) Participants with CD123+ AML (defined as ≥20% of leukemic cells expressing CD123 at any point in the course of disease)

   1. up to 3rd relapse for whom all standard or life-extending therapies have failed and for whom no potentially curative therapies are available or who are intolerant to such therapies
   2. having up to 30% blasts in a bone marrow assessment at either screening or prescreening, or having between 30% and 40% blasts for two consecutive bone marrow assessments with a minimum of one month and no more than two months apart,
   3. without hyperproliferative disease requiring cytoreductive treatment,
   4. exceptions to BM blast criterion are only possible in minor deviations in timing and/or blast count in clinically stable patients, and only with written sponsor approval. Exceptions to minimum CD123 expression are not allowed.
3. For Phase 1a escalation and Phase 1b expansion part of the trial

Participants with MRD+ AML are potentially eligible but must meet the following criteria:

1. MRD positivity must be based on assays and markers supported by consensus guidelines [Heuser2021] and in the judgment of the investigator must confer negative prognostic risk highly likely to result in relapse.
2. must have received or be ineligible for allogeneic stem cell transplant.
3. must be approved by the Sponsor for inclusion in the study. 4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. 5. Life expectancy of at least 3 months in the judgment of the investigator. 6. Adequate renal and hepatic laboratory assessments: 7. Adequate cardiac function 8. Long-term central venous access existing (e.g., port-system) or willing to have such a device inserted.

9. Able to give written informed consent. 10. Weight ≥45 kg. 11. Negative pregnancy; routinely using a highly effective method of birth control

Exclusion Criteria:

1. Acute promyelocytic leukemia (t15;17).
2. AML with only extramedullary manifestations (e.g., chloroma, primary myeloid sarcoma)
3. Acute manifestationof AML in the central nervous system.
4. Bone marrow failure syndromes
5. Cardiac disease: heart failure (New York Heart Association III or IV); unstable coronary artery disease, myocardial infarction, or serious cardiac ventricular arrhythmias requiring anti-arrhythmic therapy within the last 6 months prior to study entry.
6. Active pulmonary disease with clinically relevant hypoxia
7. Parkinson's disease or epilepsy with clinical symptoms in the previous 12 months .
8. Stroke, seizure, or intracranial hemorrhage in the past 12 months.
9. History or presence of disseminated intravascular coagulation (DIC), deep vein thrombosis or thromboembolism within 3 months prior to start of treatment.
10. Active infectious disease considered by investigator to be incompatible with protocol or being contraindications for lymphodepletion therapy
11. Presence of hemorrhagic cystitis
12. Other toxicity from prior anticancer treatment has not resolved to Grade ≤1 or baseline.
13. Allogeneic stem cell transplantation within last 2 months or GvHD requiring systemic immunosuppressive therapy.
14. Vaccination with live viruses < 2 weeks prior to lymphodepletion therapy.
15. Major surgery within 28 days prior to start of R-TM123 infusion.
16. Prior malignancy in the past 3 years or any malignancy requiring ongoing active therapy other than adjuvant endocrine therapy. Participants with resected or ablated tumors, such as basal cell carcinoma of skin, carcinoma-in-situ of the cervix, or other tumors considered cured may be considered for the study with Sponsor approval.
17. Treatment with any investigational drug substance or experimental therapy within 4 weeks or 5 half-lives (whichever is shorter) of the substance prior to lymphodepletion.
18. Treatment with anti-leukemic therapy within 4 weeks or 5 half-lives (whichever is shorter) prior to lymphodepletion.
19. Prior treatment with gene modified cell products.
20. Use of checkpoint inhibitors within 5 half-lives of the specific drug.
21. Autoimmune diseases requiring systemic steroids or other systemic immunosuppressants.
22. Pregnant or breastfeeding women.
23. Psychologic disorders with treatment modifications required within the last 3 months, drug and/or significant active alcohol abuse as per investigator's medical judgement. Depression or anxiety due to presence of the underlying malignancy may be exempted with Sponsor approval.
24. History of human immunodeficiency virus (HIV) or human T-lymphotropic virus (HTLV) or active/chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV).
25. Presence of autoantibodies against lupus La protein (La)/ Sjögren syndrome type B antigen (SS-B) or presence or history of autoimmune diseases associated with such antibodies
26. Known hypersensitivity to cellular component (Allo-RevCAR01-T) and/or TM (R-TM123) excipients or to compounds of the lymphodepletion therapy, tocilizumab, or corticosteroids.
27. Evidence that the participant is not likely or able to follow the study protocol (e.g., lacking compliance) in the judgment of the investigator.
28. Participant unable to understand the informed consent and possible consequences of the participation in the clinical trial in the judgement of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
To assess the safety profile of the treatment | At the end of cycle 1 (in total 28 days, given no treatment interruptions)
  Incidence and intensity of adverse events (AEs) graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, except for cytokine release syndrome (CRS), immune effector cell associated neurotoxicity syndrome (ICANS), tumor lysis syndrome, and graft versus host disease (GvHD), which will be graded according to widely accepted specialized criteria
To determine the incidence of dose-limiting toxicities (DLT) | At the end of cycle 1 (in total 28 days, given no treatment interruptions)
  Incidence of DLTs
To determine the maximum tolerated dose (MTD) | At the End of Cycle 1 (in total 28 days, given no treatment interruptions)
  MTD

SECONDARY OUTCOMES:
Response rate to consolidation treatment cycles | At any timepoint until end of study (6 months after the end of last R-TM123 administration)
  * Complete remission (CR, CRc, CRh, CRi, CRMRDneg, CRMRDpos)
  * Morphologic leukemia free state (MLFS),
  * Partial remission (PR)
  * Overall response rate (ORR)
  * Best response rate
  * Duration of response
Establishing recommended Phase 2 dose (RP2D) | At any timepoint until end of study (6 months after the end of last R-TM123 administration)
  Based on assessments of MTD and DLTs
Survival rates | At end of study visit (6 months after the end of last R-TM123 administration)
  * Progression free survival
  * Overall survival
Evidence of biological and clinical activity including best response rate | At any timepoint until end of study (6 months after the end of last R-TM123 administration)
  * Complete remission (CR, CRh, CRi, CRMRDneg, CRMRDpos)
  * Morphologic leukemia free state (MLFS)
  * Partial remission (PR)
  * Overall response rate (ORR)
  * Best response rate
  * Duration of response
  * PFS
  * OS

CONTACTS AND LOCATIONS:
Overall Officials: Tapan Maniar, MD, Study Director — AvenCell Europe GmbH
Locations (11):
- Germany (8):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum der Universität München, Munich, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Universitätsklinikum Marburg, Marburg, Hesse
  - Universitätsklinikum Dresden, Dresden, Saxony
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Köln, Cologne
  - Medizinische Hochschule Hannover, Hanover
- Netherlands (3):
  - Erasmus University Medical Center, Rotterdam, Gelderland
  - Amsterdam University Medical Center, Amsterdam, HV
  - University Medical Center Groningen (UMCG), Groningen, RB Groningen

IPD SHARING:
Plan to Share IPD: No